CLINICAL TRIAL: NCT06703671
Title: The Efficacy and Safety of Electroacupuncture Compared With Sham Acupuncture in Patients With Discogenic Low Back Pain: A Multicenter Randomized Controlled Trial
Brief Title: Electroacupuncture Treatment for Discogenic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Collaborators: Dongzhimen Hospital, Beijing (Other); Changshu Hospital of Traditional Chinese Medicine (Other); Shenzhen Hospital of Traditional Chinese Medicine (Unknown); First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other); Beijing Massage Hospital (Unknown); Beijing University of Chinese Medicine, Shenzhen Hospital (Other); Dongfang Hospital Beijing University of Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024BJYYEC-KY198-04; BJ-2024-205 (Other Grant/Funding Number: National High Level Hospital Clinical ResearcrFunding)
Record Dates: First submitted 2024-11-10; First posted 2024-11-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Discogenic Low Back Pain
Keywords: Discogenic low back pain; electroacupuncture; Sham Acupuncture; A Randomized Clinical Trial

STUDY DESIGN:
Intervention Model Description: In the electroacupuncture group, electroacupuncture was applied to selected acupoints for 30 min per treatment, and the treatment was performed 3 times per week (1-2 days between each treatment), receiving a total of 12 treatments in 4 weeks. Considering the possibility of uncontrollable factors such as temporary outings and overtime work during the treatment period, we will allow subjects to miss a maximum of 3 treatments, including 2 consecutive treatments.
  In the sham acupuncture group, placebo-needle treatment was performed on nonacupoints for 30 min per treatment, and the treatment was performed 3 times per week (with an interval of 1-2 days between treatments), with a total of 12 treatments received in 4 weeks. Considering the possibility of uncontrollable factors such as temporary outings, overtime work, etc. during the treatment period, we will allow subjects to miss a maximum of 3 treatments, including 2 consecutive treatments.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, outcome assessors, and statisticians were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture group (Experimental): In the electroacupuncture group, the acupuncture point prescription is based on the Evidence-based Practice Guidelines for Non-surgical Treatment of lumbar disc Herniation. The best clinical acupuncture treatment strategy was determined by the expert committee.Electroacupuncture was applied to the standard acupoints (BL-23,BL-25,EX-B2,BL-40,GB-34) for 30 min per treatment, and the treatment was performed 3 times per week (with an interval of 1-2 days between treatments), with a total of 12 treatments received over 4 weeks. Point selection and location refer to the current national standard "GB/T 12346-2021 Meridian point Name and Location".
  Interventions: Device: electroacupuncture group
- sham-acupuncture group (Sham Comparator): In the sham-acupuncture group,the prescription of this sham acupuncture scheme was made with reference to SHARE: Report Guidelines and Clinical Trial List of sham acupuncture and Research on acupuncture point Localization in the treatment of chronic low back Pain.Sham-acupuncture treatments were performed on noacupoints (Sham-BL-23,Sham-BL-25,Sham-EX-B2,Sham-BL-40,Sham-GB-34) for a duration of 30 min for each treatment session, and 3 treatments were performed per week (with an interval of 1-2 days between each treatment session), for a total of 12 treatments over 4 weeks.
  Interventions: Device: sham-acupuncture group

INTERVENTIONS:
Device: electroacupuncture group — According to the acupuncture prescription, the acupuncture doctor carried out acupuncture and lifting and twisting, and "qi" appeared under the needle. Select waist Jiaji point and Shenshu point on the same side to connect a set of electronic needle therapy instrument, the positive pole (red clip) connected to Shenshu point, the negative pole (white clip) connected to waist Jiaji point, after confirming that the electric current intensity of the electric needle instrument returns to zero, open the electronic needle therapy instrument, select continuous wave, 2Hz, current intensity 2mA. During the process of needle retention, the other points were injected every 15 minutes and retained for 30 minutes.The investigators have developed detailed acupoint positioning and operation rules.
  Arms: electroacupuncture group
Device: sham-acupuncture group — The investigators fixed the foam pad with one hand and inserted a comfort needle with the other, making sure the needle only touched the surface of the skin and did not penetrate the point. After the completion of all acupoint operations, the operator selected the simulated needle insertion points of Jiaji point on the waist and Shenshu point on the same side. An electroacupuncture treatment device designed to connect a circuit interrupt treatment is operated with the electroacupuncture group, a process that ensures that the participant does not experience any perceptible stimulation
  Arms: sham-acupuncture group

SUMMARY:
Low back pain (LBP) is a prevalent clinical condition characterized by pain localized between the lower edge of the 12th rib and the gluteal fold.The incidence of LBP has been escalating annually.An epidemiological survey encompassing 204 countries and territories globally projects a stark increase in the affected population, from an estimated 619 million in 2020 to a projected 843 million by 2050.LBP can affect individuals across all age groups, with a lifetime prevalence ranging from 60% to 80%, significantly impairing quality of life. Discogenic low back pain (DLBP), attributed to degenerative changes in the intervertebral discs, is the predominant subtype of LBP, comprising approximately 39% of all LBP cases. Disc degeneration typically initiates in early adulthood and progresses with age, potentially leading to DLBP.As the population ages, DLBP has emerged as a major contributor to disability worldwide, imposing a substantial burden on both individuals and society. Current international guidelines establish the foundation for surgical and pharmacological interventions for DLBP.However, considering the adverse effects and economic implications associated with surgical and medical treatments, there is a growing inclination towards recommending non-pharmacological therapies.These include physiotherapy, self-management, and psychotherapy, with a concurrent reduction in emphasis on pharmacological and surgical options.

Acupuncture and moxibustion are integral components of traditional Chinese medicine, garnering global recognition for their role in restoring the equilibrium of yin and yang within the human body . Electroacupuncture, a modern derivation of traditional acupuncture, has been extensively applied worldwide for the management of various painful conditions, including headache, myofibromyalgia, neck pain, and cancer-related pain. Despite its broad application, a limited number of clinical efficacy and safety studies have been conducted on electroacupuncture for the treatment of discogenic low back pain (DLBP), thereby necessitating a scientific foundation for its therapeutic use .

The present study aims to investigate the clinical efficacy and safety of electroacupuncture in the treatment of DLBP using an evidence-based medical approach. By employing a multicenter, randomized, and sham-controlled study design, this investigation seeks to provide a robust evidence-based medical foundation for the use of electroacupuncture in DLBP treatment.

Participants will be randomly assigned to either the acupuncture group (experimental group) or the sham acupuncture group (control group) in a 1:1 ratio, akin to a lottery drawing. Following enrollment, participants will undergo a 4-week, 12-session intervention, followed by three follow-up visits at 4, 12, and 24 weeks post-treatment. The investigators will assess participants' low back pain, lumbar spine function, and quality of life through telephone communication or on-site questioning at these designated follow-up intervals.

Needling may result in minor bleeding, pain, or hematoma at the needle site, and rare infections or allergic reactions may occur. Adverse reactions to needling, such as dizziness or nerve damage, are exceedingly rare.

Participants in this study may confer direct medical benefits, such as remission of symptoms, or may not, with outcomes ranging from no remission to potential exacerbation of the condition . However, the knowledge gained from this study is anticipated to benefit future people with similar conditions .

In addition to this study , participations may opt for treatment with modern rehabilitation medicine modalities or medications, including shortwave therapy, intermediate frequency therapy, or oral analgesics . This study would not impose any costs beyond the participants' regular medical treatment, and the investigators will cover all study-related medical expenses (including acupuncture treatment costs, needle costs, and scale evaluation costs) . The investigators are legally committed to maintaining the confidentiality of the participants' study records.

ELIGIBILITY:
Inclusion Criteria:

1. It meets the diagnostic criteria of discogenic low back pain
2. Betweening 18 and 70 years of age (both 18 and 70) and of either sex
3. Visual analog score (VAS) for low back pain ≥40 mm within the last 1 month

Exclusion Criteria:

1. Patients with symptoms such as lower limb numbness, weakness and claudication as shown by lumbar disc herniation pressing the spinal nerve on imaging
2. Lumbar tuberculosis, tumor, infection, spinal fracture, lumbar spondylolisthesis, severe osteoporosis
3. Patients with a history of spinal and intervertebral disc surgery
4. Patients with rheumatism, rheumatoid disease, systemic lupus erythematosus, hematopoietic system, endocrine system and psychiatric diseases
5. Patients who have received radiofrequency, minimally invasive, ozone, small needle-knife, acupuncture, manipulation, traction, block therapy and other clinical trials within the last 1 month
6. Patients with severe needle fainting intolerance
7. Women who are pregnant, planning pregnancy or breastfeeding
8. People with a history of opioid analgesics, sedatives and hypnotics and alcohol abuse
9. Patients who plan to undergo acupuncture, massage, traction and other treatments related to this disease and other clinical research trials within 3 months of participating in the study
10. Patients with skin damage or infection, concomitant bleeding tendency, tumor metastasis, serious heart disease, or embedded pacemaker

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-03-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | Measured before treatment, after 2 weeks of treatment, after 4 weeks of treatment, 4 weeks, 12 weeks and 24 weeks after the end of treatment
  Visual Analogue Scale is one of the most commonly used single-dimension measurement and evaluation tools for pain intensity. The scale is mainly composed of a 100mm straight line, one end of which means "completely painless" and the other end means "the most severe pain imaginable" or "pain to the extreme." The patient will be asked to place a mark (with a dot) on the line to represent the intensity of the pain they are experiencing at the time.A higher score means a worse result.

SECONDARY OUTCOMES:
Oswestry disability index | Measured before treatment, after 2 weeks of treatment, after 4 weeks of treatment, 4 weeks, 12 weeks and 24 weeks after the end of treatment
  The Oswestry Disability Index is a scale commonly used to assess low back pain (LBP) dysfunction. It consists of 10 questions, including pain intensity, self-care, lifting, walking, sitting, standing, sleep disturbance, social life, travel, sex life and other 10 aspects, with 6 options for each question, the highest score of each question is 5 points, 0 points for choosing the first option, and 5 points for choosing the last option in turn. If 10 questions are answered, the scoring method is: actual score /50 (highest possible score) ×100%, if a question is not answered, the scoring method is: actual score /45 (highest possible score) ×100%, if the higher indicates the more serious dysfunction.
Japanese Orthopaedic Association scores | Measured before treatment, after 2 weeks of treatment, after 4 weeks of treatment, 4 weeks, 12 weeks and 24 weeks after the end of treatment
  The Japanese Orthopaedic Association score for low back pain includes four parts: subjective symptoms (low back pain, leg pain, gait), clinical signs (straight leg lifting, sensory impairment, motor impairment), limits of daily activities and bladder function, with a total score of 29. Improvement index = post-treatment score - pre-treatment score, post-treatment score improvement rate =[(post-treatment score - pre-treatment score)/pre-treatment score]×100%. The improvement index can reflect the improvement of lumbar function before and after treatment, and the clinical treatment effect can be understood by the improvement rate. The improvement rate can also correspond to the commonly used efficacy criteria: it is a cure when the improvement rate is 100%; it is significant when the improvement rate is greater than 60%; when the improvement rate is 25%-60%, it is effective; when it is less than 25%, it is ineffective.
Hospital Anxiety and Depression Scale | Measured before treatment, after 2 weeks of treatment, after 4 weeks of treatment, 4 weeks, 12 weeks and 24 weeks after the end of treatment
  The Hospital anxiety and depression scale , which integrates the assessment of anxiety and depression, is mainly applied to the screening of anxiety and depression in patients in general hospitals, and is widely used in studies. Emotions play an important role in most illnesses, and if your doctor understands your mood changes, they can help you more. Please read the following items and put a "x" in brackets after the options that best match your mood over the past month. Don't think too much about the answers to these questions; immediate answers are often more realistic. Scoring criteria: This table includes 2 subscales of anxiety and depression, 7 questions each for anxiety [A] and depression [D].
  The subscale of anxiety and depression was divided into the following scores: 0-7 were asymptomatic; 8-10 are suspicious; The genus 11-21 definitely exists; In the scoring, the starting point is 8, that is, both suspicious and symptomatic people are positive.
the 12-items Short Form Health Survey | Measured before treatment, after 2 weeks of treatment, after 4 weeks of treatment, 4 weeks, 12 weeks and 24 weeks after the end of treatment
  The 12-item Short From Health Survey contains 12 items and 8 dimensions, which are respectively physiological function, the impact of physiological function on role function, physical pain, general health, vitality, social function, physical function. Effects of emotions on role functions, mental health.The scale was scored on a percentage scale, and the higher the score, the higher the quality of life.
Number of Participants Experiencing Adverse Reactions During Acupuncture | We will systematically monitor and document any adverse reactions (such as pain, bleeding, infection, etc.) following each session of acupuncture or sham acupuncture within a 4-week, 12-session intervention period. The observational period for this trial
  We will record the total number of participants who experience any adverse reactions (such as pain, bleeding, infection, etc.) during the acupuncture treatment.
Rate of Adverse Reactions During Acupuncture Treatment | Upon the conclusion of the trial, which is anticipated to span approximately 1.5 years, we will compute and report the incidence rate of adverse events based on the tally of occurrences.
  Following the conclusion of the study, we will determine the incidence rate of adverse reactions experienced during the course of acupuncture or sham acupuncture treatment.

OTHER OUTCOMES:
Acupuncture Treatment Expectation for Treatment Scale | Measured before the first pinprick and within 10 minutes after the last pinprick
  There are several options in the table that indicate participants' expectations for acupuncture treatment. There is no right or wrong answer. A higher score indicates a higher expectation for treatment, and a lower score indicates a lower expectation for treatment.
Acupuncture blind method implementation evaluation scale | Measured before the first pinprick and within 10 minutes after the last pinprick
  Participants in both groups were evaluated for blinding while receiving electroacupuncture or a dummy needle. Participants' feelings about the intervention were recorded with "yes," "no," or "unclear."

CONTACTS AND LOCATIONS:
Overall Officials: Guodong Ni, MMed, Study Chair — Department of Acupuncture and Massage, Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data with others for six months after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD analysis will be shared by June 1, 2026.
Access Criteria: The data shared will include participant characteristics, clinical measurements, adverse events, and clinical outcomes. This data will be provided through a secure online platform or database, ensuring data security and privacy protection. The data will be shared with researchers who make legitimate requests for data, including research hypotheses, research justifications, analysis plans, publication plans, and the credentials of the research team.

REFERENCES:
- [Result] Lee B, Kwon CY, Lee HW, Nielsen A, Wieland LS, Kim TH, Birch S, Alraek T, Lee MS. Needling Point Location Used in Sham Acupuncture for Chronic Nonspecific Low Back Pain: A Systematic Review and Network Meta-Analysis. JAMA Netw Open. 2023 Sep 5;6(9):e2332452. doi: 10.1001/jamanetworkopen.2023.32452. PMID 37672270
- [Result] Ma P, Liu X, Liu Z, Guo Y, Zhou K, Bian Z, Sun C, Liu T, Xiong Z, Xie Y, Lu Y, Lao L, He L, Liu B, Liu C, Yan S; SHARE Workgroup. The SHARE: SHam Acupuncture REporting guidelines and a checklist in clinical trials. J Evid Based Med. 2023 Dec;16(4):428-431. doi: 10.1111/jebm.12560. Epub 2023 Oct 31. No abstract available. PMID 37906211
- [Result] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Result] Tu JF, Shi GX, Yan SY, Ni GX, Yu FT, Cai GW, Liu ZS, Ma CY, Wang LQ, Yang JW, Zhou XQ, Meng XL, Fu HY, Li J, Wan WJ, Sun TH, Wang XZ, Liu CZ. Acupuncture vs Sham Acupuncture for Chronic Sciatica From Herniated Disk: A Randomized Clinical Trial. JAMA Intern Med. 2024 Dec 1;184(12):1417-1424. doi: 10.1001/jamainternmed.2024.5463. PMID 39401008
- [Result] Kreiner DS, Matz P, Bono CM, Cho CH, Easa JE, Ghiselli G, Ghogawala Z, Reitman CA, Resnick DK, Watters WC 3rd, Annaswamy TM, Baisden J, Bartynski WS, Bess S, Brewer RP, Cassidy RC, Cheng DS, Christie SD, Chutkan NB, Cohen BA, Dagenais S, Enix DE, Dougherty P, Golish SR, Gulur P, Hwang SW, Kilincer C, King JA, Lipson AC, Lisi AJ, Meagher RJ, O'Toole JE, Park P, Pekmezci M, Perry DR, Prasad R, Provenzano DA, Radcliff KE, Rahmathulla G, Reinsel TE, Rich RL Jr, Robbins DS, Rosolowski KA, Sembrano JN, Sharma AK, Stout AA, Taleghani CK, Tauzell RA, Trammell T, Vorobeychik Y, Yahiro AM. Guideline summary review: an evidence-based clinical guideline for the diagnosis and treatment of low back pain. Spine J. 2020 Jul;20(7):998-1024. doi: 10.1016/j.spinee.2020.04.006. Epub 2020 Apr 22. PMID 32333996
- [Result] Kim G, Kim D, Moon H, Yoon DE, Lee S, Ko SJ, Kim B, Chae Y, Lee IS. Acupuncture and Acupoints for Low Back Pain: Systematic Review and Meta-Analysis. Am J Chin Med. 2023;51(2):223-247. doi: 10.1142/S0192415X23500131. Epub 2022 Dec 31. PMID 36585839
- [Result] He Y, Guo X, May BH, Zhang AL, Liu Y, Lu C, Mao JJ, Xue CC, Zhang H. Clinical Evidence for Association of Acupuncture and Acupressure With Improved Cancer Pain: A Systematic Review and Meta-Analysis. JAMA Oncol. 2020 Feb 1;6(2):271-278. doi: 10.1001/jamaoncol.2019.5233. PMID 31855257
- [Result] Castellini G, Pillastrini P, Vanti C, Bargeri S, Giagio S, Bordignon E, Fasciani F, Marzioni F, Innocenti T, Chiarotto A, Gianola S, Bertozzi L. Some conservative interventions are more effective than others for people with chronic non-specific neck pain: a systematic review and network meta-analysis. J Physiother. 2022 Oct;68(4):244-254. doi: 10.1016/j.jphys.2022.09.007. Epub 2022 Oct 17. PMID 36266185
- [Result] Deare JC, Zheng Z, Xue CC, Liu JP, Shang J, Scott SW, Littlejohn G. Acupuncture for treating fibromyalgia. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD007070. doi: 10.1002/14651858.CD007070.pub2. PMID 23728665
- [Result] Coeytaux RR, Befus D. Role of Acupuncture in the Treatment or Prevention of Migraine, Tension-Type Headache, or Chronic Headache Disorders. Headache. 2016 Jul;56(7):1238-40. doi: 10.1111/head.12857. Epub 2016 Jul 13. PMID 27411557
- [Result] Chen HY, Yeung WF, Yang MX, Mu JL, Ziea TC, Ng Bacon FL, Lao LX. Guideline Acupuncture for low back pain: a clinical practice guideline from the Hong Kong taskforce of standardized acupuncture practice. J Tradit Chin Med. 2022 Feb;42(1):140-147. doi: 10.19852/j.cnki.jtcm.2022.01.009. PMID 35294134
- [Result] Tang X, Shi X, Zhao H, Lu L, Chen Z, Feng Y, Liu L, Duan R, Zhang P, Xu Y, Cui S, Gong F, Fei J, Xu NG, Jing X, Guyatt G, Zhang YQ. Characteristics and quality of clinical practice guidelines addressing acupuncture interventions: a systematic survey of 133 guidelines and 433 acupuncture recommendations. BMJ Open. 2022 Feb 24;12(2):e058834. doi: 10.1136/bmjopen-2021-058834. PMID 35210347
- [Result] Foster NE, Anema JR, Cherkin D, Chou R, Cohen SP, Gross DP, Ferreira PH, Fritz JM, Koes BW, Peul W, Turner JA, Maher CG; Lancet Low Back Pain Series Working Group. Prevention and treatment of low back pain: evidence, challenges, and promising directions. Lancet. 2018 Jun 9;391(10137):2368-2383. doi: 10.1016/S0140-6736(18)30489-6. Epub 2018 Mar 21. PMID 29573872
- [Result] Nicol V, Verdaguer C, Daste C, Bisseriex H, Lapeyre E, Lefevre-Colau MM, Rannou F, Roren A, Facione J, Nguyen C. Chronic Low Back Pain: A Narrative Review of Recent International Guidelines for Diagnosis and Conservative Treatment. J Clin Med. 2023 Feb 20;12(4):1685. doi: 10.3390/jcm12041685. PMID 36836220
- [Result] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Result] Sakai D, Nakamura Y, Nakai T, Mishima T, Kato S, Grad S, Alini M, Risbud MV, Chan D, Cheah KS, Yamamura K, Masuda K, Okano H, Ando K, Mochida J. Exhaustion of nucleus pulposus progenitor cells with ageing and degeneration of the intervertebral disc. Nat Commun. 2012;3:1264. doi: 10.1038/ncomms2226. PMID 23232394
- [Result] Zhang YG, Guo TM, Guo X, Wu SX. Clinical diagnosis for discogenic low back pain. Int J Biol Sci. 2009 Oct 13;5(7):647-58. doi: 10.7150/ijbs.5.647. PMID 19847321
- [Result] Fujii K, Yamazaki M, Kang JD, Risbud MV, Cho SK, Qureshi SA, Hecht AC, Iatridis JC. Discogenic Back Pain: Literature Review of Definition, Diagnosis, and Treatment. JBMR Plus. 2019 Mar 4;3(5):e10180. doi: 10.1002/jbm4.10180. eCollection 2019 May. PMID 31131347
- [Result] Ohtori S, Inoue G, Miyagi M, Takahashi K. Pathomechanisms of discogenic low back pain in humans and animal models. Spine J. 2015 Jun 1;15(6):1347-55. doi: 10.1016/j.spinee.2013.07.490. Epub 2014 Mar 20. PMID 24657737
- [Result] GBD 2021 Low Back Pain Collaborators. Global, regional, and national burden of low back pain, 1990-2020, its attributable risk factors, and projections to 2050: a systematic analysis of the Global Burden of Disease Study 2021. Lancet Rheumatol. 2023 May 22;5(6):e316-e329. doi: 10.1016/S2665-9913(23)00098-X. eCollection 2023 Jun. PMID 37273833
- [Result] Dionne CE, Dunn KM, Croft PR, Nachemson AL, Buchbinder R, Walker BF, Wyatt M, Cassidy JD, Rossignol M, Leboeuf-Yde C, Hartvigsen J, Leino-Arjas P, Latza U, Reis S, Gil Del Real MT, Kovacs FM, Oberg B, Cedraschi C, Bouter LM, Koes BW, Picavet HS, van Tulder MW, Burton K, Foster NE, Macfarlane GJ, Thomas E, Underwood M, Waddell G, Shekelle P, Volinn E, Von Korff M. A consensus approach toward the standardization of back pain definitions for use in prevalence studies. Spine (Phila Pa 1976). 2008 Jan 1;33(1):95-103. doi: 10.1097/BRS.0b013e31815e7f94. PMID 18165754